CLINICAL TRIAL: NCT01870245
Title: A Phase 1 Multiple Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of ACHN-975 Administered Intravenously to Healthy Volunteers
Brief Title: A Multiple Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of ACHN-975 in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Achaogen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACHN-975-002
Record Dates: First submitted 2013-05-29; First posted 2013-06-06 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — ACHN-975

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ACHN-975 (Experimental)
  Interventions: Drug: ACHN-975
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ACHN-975 — Intravenous multiple dose
  Arms: ACHN-975
Drug: placebo — Intravenous multiple dose
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multiple-dose study, designed to assess the safety, tolerability, and pharmacokinetics (PK) of ACHN-975. This study will take place in the US at one clinical site.

ELIGIBILITY:
Key Inclusion Criteria:

* Body weight between 40 and 100 kilograms (between ~88 pounds and ~220 pounds)
* Use of contraception
* Stable health
* Negative tests for alcohol, tobacco, and drugs of abuse

Key Exclusion Criteria:

* History of clinically significant disease
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Frequency of AEs | 28 days
Severity of AEs | 28 days

SECONDARY OUTCOMES:
Plasma concentrations of ACHN-975 | 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Achaogen, Inc.
Locations (1):
- Investigational Site, Overland Park, Kansas, United States